CLINICAL TRIAL: NCT06884904
Title: Umbilical Mesenchymal Stem Cells in the Treatment of Acute-on-Chronic Liver Failure：A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase IIb/III Seamless Adaptive Design Clinical Study
Brief Title: Umbilical Cord-derived Mesenchymal Stem Cell Infusion for Treating ACLF
Acronym: MSCTACLF
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Engineering Center of Cell Products (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSCTACLF-02
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Acute-On-Chronic Liver Failure
Keywords: acute-on-chronic liver failure; mesenchymal stem cells
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low-dose experimental group (Experimental): 2.0×10^6/kg
  Interventions: Drug: Low-dose experimental group
- High-dose experimental group (Experimental): 4.0×10^6/kg
  Interventions: Drug: High-dose experimental group
- Low-dose placebo control group (Placebo Comparator): Equivalent volume of solvent calculated at 2.0×10^6/kg
  Interventions: Drug: Low-dose placebo control group
- High-dose placebo control group (Placebo Comparator): Equivalent volume of solvent calculated at 4.0×10^6/kg
  Interventions: Drug: High-dose placebo control group

INTERVENTIONS:
Drug: Low-dose experimental group — 2.0*10^6/kg
  Arms: Low-dose experimental group
Drug: High-dose experimental group — 4.0*10^6/kg
  Arms: High-dose experimental group
Drug: Low-dose placebo control group — Equivalent volume of solvent calculated at 2.0×10^6/kg
  Arms: Low-dose placebo control group
Drug: High-dose placebo control group — Equivalent volume of solvent calculated at 4.0×10^6/kg
  Arms: High-dose placebo control group

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled adaptive design Phase IIb/III clinical trial. It employs a seamless adaptive design, divided into Phase IIb and Phase III, focusing on patients with acute-on-chronic liver failure (ACLF). Eligible patients meeting the inclusion criteria and not disqualified were randomized in a 2:2:1:1 ratio during Phase IIb to receive either a high-dose experimental group (4.0×10^6/kg of injectable mesenchymal stem cells derived from umbilical cord), a low-dose group (2.0×10^6/kg), a high-dose placebo control group (with equivalent volume of solvent calculated at 4.0×10^6/kg), or a low-dose placebo control group (with equivalent volume of solvent calculated at 2.0×10^6/kg). In Phase III, patients were randomized in a 1:1 ratio to the experimental group (injectable umbilical cord-derived mesenchymal stem cells) or the control group. All groups received standard treatment alongside either the experimental drug (experimental group) or placebo (control group) to evaluate and confirm the efficacy and safety of injectable umbilical cord-derived mesenchymal stem cells in treating acute-on-chronic liver failure.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years (inclusive) at the time of signing the informed consent form, regardless of gender.
2. Patients with hepatitis B virus (HBV)-associated acute-on-chronic liver failure (ACLF) meeting the following criteria: Total bilirubin (TBil) ≥12 mg/dL (equivalent to 205 μmol/L); International normalized ratio (INR) ≥1.5 or prothrombin activity (PTA) ≤40%;
3. All participants and their partners agree to use effective non-pharmacological contraception during the trial and for 6 months after trial completion, with no plans for conception during this period.
4. Voluntarily participate in the clinical study and sign the informed consent form.

Exclusion Criteria:

1. History of allergy to any component of the investigational drug or bovine-derived products.
2. Acute, subacute, or chronic liver failure unrelated to HBV, or ACLF caused by: Concurrent hepatitis A, C, or E virus infection; Autoimmune liver disease; Biliary obstruction.
3. Presence of any of the following complications: <1> Active gastrointestinal bleeding (e.g., hematemesis and/or melena) or high- risk esophageal/gastric varices (confirmed by endoscopy or imaging within 3 months prior to screening). <2> Imaging evidence (ultrasound or CT) of cavernous transformation of the portal vein or portal vein occlusion. <3> History of transjugular intrahepatic portosystemic shunt (TIPS). <4> Grade 3 or 4 hepatic encephalopathy. <5> Serum creatinine ≥2 mg/dL. <6> Respiratory insufficiency (e.g., dyspnea, cyanosis) with peripheral oxygen saturation ≤93% at rest.
4. Severe underlying diseases, including: <1>Septic shock (requiring vasopressors to maintain mean arterial pressure ≥65 mmHg despite adequate fluid resuscitation, with blood lactate >2 mmol/L). <2> Uncontrolled cardiac conditions: Myocardial ischemia or infarction (CTCAE v5.0 Grade ≥II), Arrhythmias requiring intervention, NYHA Class III-IV heart failure. <3> Active malignancy (solid or hematologic). <4> Diagnosed pulmonary hypertension or suspected pulmonary embolism. <5> IgA deficiency, Henoch-Schönlein purpura, hemophilia, or idiopathic thrombocytopenia. <6> Immunodeficiency disorders (e.g., HIV infection, congenital/acquired immune deficiency).
5. Current systemic corticosteroid therapy for other diseases.
6. Psychiatric or other conditions deemed by the investigator to interfere with study assessments.
7. Planned or active registration for liver transplantation, or anticipated transplantation within 3 months.
8. History of liver transplantation.
9. Alcohol or substance abuse: Chronic alcohol use (>5 years with ethanol intake ≥40 g/day for males or ≥20 g/day for females), Heavy alcohol use (>80 g/day ethanol) within 2 weeks prior to screening, Abstinence <6 months.
10. Participation in another clinical trial within 3 months prior to screening (excluding screen failures or withdrawal before dosing).
11. Pregnancy, lactation, or positive pregnancy test at screening.
12. Any other condition that, in the investigator's judgment, may confound study results, pose risks, or compromise the participant's best interests.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-04-14 (Estimated); Study Completion 2028-04-14 (Estimated)

PRIMARY OUTCOMES:
mortality rate | 90 day
  90 day mortality rate (D90) of subjects randomly assigned and receiving the investigational drug

IPD SHARING:
Plan to Share IPD: No